# **COVER PAGE**

| Official Title: | A Phase 3b/4 Randomized, Double-Blind, Placebo-Controlled, Parallel- Group Study to Verify the Clinical Benefit of Aducanumab (BIIB037) in Participants with Alzheimer's Disease |
|---|---|
| NCT Number: | NCT05310071 |
| Document Date: | 06 May 2024 |

Product: Aducanumab
Study: 221AD305
Statistical Analysis Plan
Version: 1.0



# STATISTICAL ANALYSIS PLAN

Version No.: 1.0

Date: 6 May 2024

Author:

Study Title: A Phase 3b/4 Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Verify the Clinical Benefit of Aducanumab (BIIB037) in Participants with Alzheimer's Disease

Name of Study Treatment: Aducanumab

Protocol No.: 221AD305

Study Phase: 3b/4

#### **Confidential Information**

The information contained in this Statistical Analysis Plan (SAP) is confidential and may not be reproduced or otherwise disseminated without the approval of Biogen, Inc.

Product: Aducanumab
Study: 221AD305
Statistical Analysis Plan
Version: 1.0

# **APPROVAL**



Product: AducanumabStatistical Analysis PlanStudy: 221AD305Version: 1.0

# **VERSION HISTORY**

| SAP Version | Date | Primary Reasons for<br>Amendment |
|-------------|------------|----------------------------------|
| V1.0 | 6 May 2024 | Not applicable |

Product: AducanumabStatistical Analysis PlanStudy: 221AD305Version: 1.0

# **TABLE OF CONTENTS**

| ST. | ATISTI | CAL ANALYSIS PLAN | 1 |
|---|---|---|---|
| ΑP | PROVA | <b>XL</b> | 2 |
| VE | RSION | HISTORY | 3 |
| TA | BLE O | F CONTENTS | 4 |
| LIS | ST OF T | ABLES Error! Bookmark not | t defined |
| LIS | ST OF A | ABBREVIATIONS | 7 |
| 1. | | Introduction | 10 |
| 2. | 2.1. | Study Overview | 11<br>11 |
| | 2.1.1. | Tertiary Objectives and Endpoints Related to Safety and Immunogenicity | 11 |
| | 2.2. | Study Design | 11 |
| | 2.2.1. | Study Overview | 11 |
| | 2.2.2. | Substudies | 13 |
| | 2.2.3. | Study Conduct Following Announcement of Study Termination | 13 |
| | 2.2.4.<br>Termi | Procedures for Releasing Treatment Assignments Following Announcement of St | • |
| | 2.2.5. | Changes to Study Execution Following Announcement of Study Termination | 13 |
| | 2.2.6. | Sample Size Considerations | 15 |
| 3. | 3.1. | Definitions Dates and Points of Reference | |
| | 3.2. | Study Treatment | 18 |
| | 3.3. | Study Periods | 18 |
| | 3.4. | Key Derived Variables | 19 |
| | 3.4.1. | Composite Score Derivation of CDR Subscores and CDR Global Score | 19 |
| | 3.5. | Stratification Factors | 19 |
| | 3.6. | Analysis Sets | 19 |
| | 3.6.1. | Randomized Set | 19 |
| | 3.6.2. | Full Analysis Set (FAS) | 19 |
| | 3.6.3. | Safety Analysis Set | 19 |
| | 3.6.4. | Safety MRI Analysis Set | 19 |
| | 3.6.5. | Immunogenicity Analysis Set | 20 |

| 4. | 4.1. | List of Planned Study Analyses Interim Analysis | |
|---|---|---|---|
| | 4.2. | Primary Analysis | 21 |
| | 4.3. | Final Analysis | 21 |
| 5. | 5.1. | Statistical Methods for Planned Analyses General Principles | |
| | 5.1.1. | High Level Description of Analyses | 22 |
| | 5.1.2. | Handling of Missing Data on Clinical Measures | 22 |
| | 5.2. | Participant Accountability | 23 |
| | 5.3. | Demographic and Baseline Characteristics | 23 |
| | 5.4. | Protocol Deviations | 23 |
| | 5.5. | Study Treatment Exposure and Concomitant Medications | 24 |
| | 5.5.1. | Study Drug Exposure and Study Drug Compliance | 24 |
| | 5.5.2. | Concomitant Medications | 24 |
| | 5.6. | Efficacy Endpoints | 25 |
| | 5.7. | Safety Endpoints | 25 |
| | 5.7.1. | Adverse Events | 25 |
| | 5.7.2. | Clinical Laboratory Evaluations | 30 |
| | 5.7.3. | Vital Signs | 32 |
| | 5.7.4. | Physical Examination and Neurological Examination | 32 |
| | 5.7.5. | Electrocardiograms | 32 |
| | 5.7.6. | Immunogenicity | 33 |
| | 5.7.7. | C-SSRS | 34 |
| 6. | 6.1. | Changes from Protocol-Specified Analyses | |
| | 6.2. | Tertiary Endpoints | 35 |
| | | | 35 |
| 7. | | Summary of Changes from the Previous Version of the SAP | 36 |
| 8. | | References | 37 |
| 9. | 9.1. | Appendix | |
| | 9.1.1. | Visit Windows for Mapping Efficacy Endpoint CDR-SB | 38 |
| | 9.1.2. | Visit Windows for Mapping Laboratory Parameters | 39 |
| | 9.1.3. | Visit Windows for Mapping Vital Sign Parameters | 39 |

| Product: Aducanumab<br>Study: 221AD305 | | Statistical Analysis Plan<br>Version: 1.0 |
|---|---|---|
| 9.1.4. | Visit Windows for Mapping Immunogenicity | 41 |
| 9.1.5. | Visit Windows for Mapping Brain MRI | 42 |
| 9.2. | Protocol Deviation Classification | 42 |
| LIST OF | TABLES | |
| Table 1<br>Visit for the | Revised Schedule of Activities for Early Termination Visit and Formula Terminated ENVISION Study | _ |
| Table 2 | Planned Analyses of all AEs, most frequent reported AEs, related 26 | AEs, and AEs by severity. |
| Table 3 | Analyses of Incidence Proportion for SAE | 27 |
| Table 4 | Verbatim Terms and MedDRA Preferred Terms | 27 |
| Table 5 | Analyses to Describe Incidence of AESIs and to Characterize AES | I Events29 |
| Table 6 | Visit Windows for Efficacy Endpoint CDR-SB | 39 |
| Table 7 | Visit Windows for Laboratory Parameters | 39 |
| Table 8 | Visit Windows for Vital Sign Parameters | 39 |
| Table 9 | Visit Windows for Immunogenicity | 41 |
| Table 10 | Visit Window for Brain MRI | 42 |
| Table 11 | Summary of Protocol Deviation Classification | 42 |
| LIST OF | FIGURES | |
| Figure 1 | Study Design Schematic | 12 |

# LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| Abs | antibodies |
| AD | Alzheimer's disease |
| ADA | Anti-drug antibodies |
| ADAS-Cog13 | Alzheimer's Disease Assessment Scale-Cognitive Subscale (13 items) |
| ADCS-ADL-MCI | Alzheimer's Disease Cooperative Study-Activities of Daily Living<br>Inventory (Mild Cognitive Impairment version) |
| AE | adverse event |
| AESI | adverse event of special interest |
| ALT | alanine aminotransferase |
| ApoE | apolipoprotein E |
| ARIA | amyloid related imaging abnormalities |
| ARIA-E | amyloid-related imaging abnormality-edema |
| ARIA-H | amyloid-related imaging abnormality-hemorrhage |
| AST | aspartate aminotransferase |
| BMI | body mass index |
| BL | baseline |
| CDR | Clinical Dementia Rating |
| CDR-SB | Clinical Dementia Rating-Sum of Boxes |
| COVID-19 | coronavirus disease 2019 |
| CNS | central nervous system |
| CRF | case report form |
| CSF | cerebrospinal fluid |
| CSR | clinical study report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| DHA | Directions for handling and administration |
| DSF | Diagnostic staging form |
| | st |
| ECG | electrocardiogram |

| Abbreviation | Definition |
|---|---|
| EDC | electronic data capture |
| EOS | end of study |
| EOT | end of treatment |
| EMACC | Early Alzheimer's Disease/Mild Cognitive Impairment Alzheimer's Cognitive Composite |
| EQ-5D-5L | health-related EuroQoL 5-dimension instrument |
| ET | early termination |
| FA | final analysis |
| FAS | full analysis set |
| FDA | Food and Drug Administration |
| FU | follow-up |
| GST | Global statistical test |
| HEOR | Health economic and outcomes research |
| HLT | high level term |
| IA | interim analysis |
| iADRS | Integrated Alzheimer's Disease Rating Scale |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IDMC | independent data monitoring committee |
| IRB | Institutional Review Board |
| IRT | interactive response technology |
| IV | intravenous |
| IXRS | Interactive Voice/Web Response System |
| LAR | Legal Authorized Representative |
| MCI | mild cognitive impairment |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMSE | Mini-Mental State Examination |
| MRI | magnetic resonance imaging |
| NIA-AA | National Institute on Aging-Alzheimer's Association |
| NPI-10 | Neuropsychiatric Inventory-10 |

| Abbreviation | Definition |
|---|---|
| PA | primary analysis |
| PC | placebo-control |
| PCS | potentially clinically significant |
| PD | pharmacodynamic(s) |
| PET | positron emission tomography |
| PK | pharmacokinetic(s) |
| PT | preferred term |
| PV4 | protocol version 4 |
| Q4W | every 4 weeks |
| QoL | quality of life |
| QoL-AD | Quality of Life in Alzheimer's Disease |
| RBANS | Repeatable Battery for the Assessment of Neuropsychological Disease Severity |
| RDV | Research Diagnostic Verification |
| RUD-Lite | Resource Utilization in Dementia – Lite Version |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SM | Site Monitor |
| SMQ | standardized MedDRA query |
| SOC | system organ class |
| SUVR | standardized uptake value ratio |
| TMA | Therapeutic Medical Advisor |
| UB | Unblinded |
| ULN | Upper limit of normal |
| WHO | World Health Organization |

#### 1. Introduction

Study 221AD305, also called the ENVISION study, was designed as a Phase 3b/4 randomized, double-blind, placebo-controlled, parallel-group study to verify the clinical benefit of aducanumab (BIIB037) in participants with Alzheimer's disease (AD). The primary study objective was to verify the clinical benefit of monthly doses of aducanumab on Clinical Dementia Rating Sum of Boxes (CDR-SB) relative to placebo at Week 78. The total duration of the study for each participant was planned to be approximately 130 weeks, including a series of screening visits within 8 weeks before administration of the first dose of study treatment, and a 104-week placebo-controlled treatment period followed by a safety follow-up (FU) visit 18 weeks after the final dose of study treatment.

Participants were scheduled to receive IV infusions of aducanumab or placebo approximately Q4W for 104 weeks. Participants were randomized to receive aducanumab: placebo in a 2:1 ratio. Aducanumab was initiated with a 6-dose titration period prior to reaching the target dose of 10 mg/kg.

Early termination of the study was announced on 31 January 2024. The decision was not related to any safety or efficacy concerns. Enrollment in 221AD305 was halted immediately upon the announcement. As a result, the planned primary analysis and optional interim analysis that were outlined in the 221AD305 protocol version 2.0, dated 15 April 2022, will not be conducted. Biogen offered the study participants the option to continue to receive treatment in a blinded fashion until 1 May 2024 to allow study participants and their health care providers sufficient time to plan future treatment decisions. Study participants were required to perform an early termination (ET) visit within 30 days of their last dose and a safety FU visit 12 weeks after their last dose. Due to the early termination of the study, an abbreviated clinical study report is planned.

The purpose of this SAP is to delineate the analyses that are planned for the final report. The primary endpoint, key secondary endpoints, and secondary endpoints of the study will not be evaluable due to the small sample size at the primary timepoint of Week 78 and key timepoints of Week 104 and Week 106. Instead, the focus of the final analysis will be summarizing the available safety data that were collected during the study to the full extent, and summarizing the available disposition, baseline characteristics, demographics, exposure, and protocol deviation data. In addition, the primary endpoint CDR-SB will be summarized by visit.

## 2. Study Overview

#### 2.1. Study Objectives and Endpoints

As mentioned in Section 1, the primary endpoint, key secondary endpoints, and secondary endpoints of the study will not be evaluable due to the small sample size at the primary timepoint of Week 78. Instead, the focus of the final analysis will be to summarize the full safety data and the data on disposition, baseline characteristics, demographics, exposure, and protocol deviations that were collected during the study. The primary endpoint CDR-SB will also be summarized by visit.

As a result, the tertiary study objectives and endpoints related to safety and immunogenicity will be the only study objectives and endpoints to be described in this section.

# 2.1.1. Tertiary Objectives and Endpoints Related to Safety and Immunogenicity

- · To assess the safety of monthly doses of aducanumab
  - Incidence of AEs and SAEs
  - o Incidence of ARIA-E and ARIA-H
  - Clinical laboratory shifts in reported values
- To assess the immunogenicity of aducanumab
  - o Incidence of anti-aducanumab antibodies (Abs) in serum over time

#### 2.2. Study Design

#### 2.2.1. Study Overview

Study 221AD305 is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study in participants with early Alzheimer's disease, including those with MCI due to Alzheimer's disease or mild Alzheimer's disease dementia. Enrollment will be monitored, via the IRT system, so that the population of participants with mild Alzheimer's disease represents approximately 50% of the total number of participants enrolled in the study. The study will include up to 24 months of treatment as well as screening and post-treatment FU periods. Approximately 1512 participants will be enrolled across an estimated 220 centers globally.

The primary study objective is to verify the clinical benefit of monthly doses of aducanumab on CDR-SB relative to placebo at Week 78. Key secondary objectives include assessment of the effect of monthly doses of aducanumab on clinical decline as compared to placebo at Week 78 as measured by a variety of cognitive and functional scales such as those implemented in the Phase 3 studies (i.e., ADCS-ADL-MCI, ADAS-Cog13, MMSE, and NPI-10), as well as the composite scale, iADRS, which is a linear combination of the ADAS-Cog13 and the ADCS-ADL-MCI. Secondary objectives include assessment of the effect of monthly doses of aducanumab on change in amyloid PET and tau PET signal at Week 78 and 104 as compared with placebo, as well as all clinical endpoints (i.e., CDR-SB, iADRS, ADCS-ADL-MCI, ADAS-Cog13, MMSE, and NPI-10) assessed at the Week 106 timepoint. Secondary objectives also include an assessment of the effect of monthly doses of aducanumab on the GST composite z-score, defined as the average of standardized z scores of the CDR-SB, ADCS-ADL-MCI, and ADAS-Cog13, at Weeks 78 and 106. Tertiary objectives include confirmation of the safety, tolerability, and associated immunogenicity of aducanumab and its PK characteristics, and HEOR and QoL metrics.

Participants will receive IV infusions of aducanumab or placebo approximately Q4W for 104 weeks. Participants will be randomized to receive aducanumab or placebo in a 2:1 ratio. The randomization will be stratified by geographical region, baseline disease stage (MCI due to Alzheimer's disease or mild Alzheimer's disease dementia), and ApoE &4 status (carrier or noncarrier). Randomization will be performed using IRT. Aducanumab will be initiated with a 6-dose titration period prior to reaching the target dose of 10 mg/kg, as detailed in Protocol Section 3.1.2 and Figure 1.

Investigators, outcome assessors, study site staff (except for the designated unblinded pharmacist/technician), study participants, and informants will be blinded to the randomized treatment assignment.

In the original study design per protocol, the total duration of the study for each participant was approximately 130 weeks, including a series of screening visits within 8 weeks before administration of the first dose, and a 104-week placebo-controlled treatment period. Participants were additionally planned to undergo a safety FU visit 18 weeks after the final dose of aducanumab.

See Figure 1 for originally planned schematic of the study design per protocol.

For schedule of activities, see Protocol Section 1.3.

Figure 1 Study Design Schematic



#### 2.2.2. Substudies

In the original study design per protocol, three optional longitudinal substudies were planned to be completed within this study in subsets of consenting participants, as follows:

- An amyloid PET substudy involving assessments of amyloid by PET scan at Screening and at Weeks 78 and 104
- A tau PET substudy involving assessments of tau by PET scan at Screening and at Weeks 78 and 104

For participants of these studies, study-specific procedures were required for provision of baseline PET scans

## 2.2.3. Study Conduct Following Announcement of Study Termination

On 31 January 2024, Biogen announced the early termination of Study 221AD305. The decision was not related to any safety or efficacy concerns. Enrollment in 221AD305 was halted immediately upon the announcement. At that time, over 1000 participants had been enrolled in the study.

Following early termination of the study, Biogen offered the study participants the option to continue to receive treatment in a blinded fashion until 1 May 2024 to allow study participants and their health care providers sufficient time to plan future treatment decisions.

# 2.2.4. Procedures for Releasing Treatment Assignments Following Announcement of Study Termination

As described in 221AD305 unblinding plan version 3.4, Biogen also decided to provide the treatment assignment information to the investigators, site staff and study participants in a patient-centric fashion, such that all study participants' treatment assignments are planned to be released to the investigators and designated site staff after the date of last patient last dose and prior to the date of the final database lock. In the event that a study participant is not interested in continuing treatment within the study until 1 May 2024 and decides to request the treatment assignment release prior to the date of last patient last dose, Biogen agreed to release treatment assignment to the corresponding investigator and the designated site staff following such requests. Blinded Biogen/IQVIA study team members will remain blinded and will not have access to the subject treatment assignments until final database lock.

#### 2.2.5. Changes to Study Execution Following Announcement of Study Termination

1) On 31 January 2024, it was announced that as the study is early terminated, participants enrolled in the study may continue receiving treatment until 01 May 2024. Screening and enrollment would be closed for the study. The participant and care partner, as applicable, should return to the site for a safety follow-up visit 30 days after their last dose. On 16 February 2024, Biogen released a document 221AD305 ENVISION Clarification Letter\_16FEB2024\_Final Signed, which updated the changes to study execution: Early Termination Visit: assessments and timing (Protocol Section 1.3, Table 2)

Due to the early termination of the study, all participants will be asked to complete this early termination (ET) visit, which, to reduce participant burden, will be limited to assessments related

to participant safety. These assessments are reported in Table 1. Participants should complete this ET visit within 30 days of their last dose of study treatment.

2) Follow-up/End of Study (FU/EOS) Visit: assessments and timing (Protocol Section 1.3, Table 2)

Due to the early termination of the study, all participants are asked to complete their Follow-up/End of Study visit (also referred to as the safety follow-up visit) at 12 weeks (+/- 3 days) after the participant's last dose of study treatment. Participants who wish to withdraw and not receive additional dosing through 01 May 2024 are still encouraged to have a safety follow-up visit 12 weeks from their last dose of study treatment. In addition, similar to the ET visit, the number of assessments that need to be completed is now reduced to lessen participant burden. These assessments are reported below in Table 1. If a participant has had their last dose of study treatment and it has been more than 12 weeks since their last dose and the participant has not had their safety follow-up, then they should complete a safety follow-up visit within 30 days, as defined in Table 1.

3) Substudies (Protocol Section 5.1)

Due to the early termination of the study, all the longitudinal substudies are terminated and samples will no longer be collected for amyloid PET, tau PET, at Weeks 52, 78, and 104/ET.

4) Management of participants who had already discontinued treatment and who were following the visit schedule defined in Table 3 (Protocol Section 1.3, Table 3)

Due to the early termination of the study, participants who discontinued treatment but agreed to remain in the study and follow the abbreviated visit schedule will be asked to complete their ET visit within 30 days and their FU/EOS visit (safety follow-up) visit 12 weeks after their last dose. If they have already had an ET visit following their last dose of treatment, then the ET visit does not need to be repeated. If it has been more than 12 weeks since their last dose and the participant has not had their safety follow-up, then they should complete a safety follow-up visit within 30 days, as defined in Table 1.

5) Visits at Week 26, Week 50, and unscheduled for Change in AD Meds (Protocol Section 1.3, Table 1 and Table 2)

Due to the discontinuation of the Aduhelm program and the early termination of the study, the visits at Week 26, Week 50, and unscheduled for change in AD medication will no longer need to be conducted as only clinical efficacy assessments are collected at these visits.

Table 1 Revised Schedule of Activities for Early Termination Visit and Followup/End of Study Visit for the Terminated ENVISION Study

| Study Assessments <sup>1</sup> | Early Termination Visit (within 30 days of last dose) | Follow up/End of Study<br>Visit <sup>2,3</sup> (12 weeks after last<br>dose +/- 3 days) |
|---|---|---|
| Body Weight | X | X |
| Urine Pregnancy Test <sup>4</sup> | X | X |

| Study Assessments <sup>1</sup> | Early Termination Visit (within 30 days of last dose) | Follow up/End of Study<br>Visit <sup>2,3</sup> (12 weeks after last<br>dose +/- 3 days) |
|---|---|---|
| Physical Exam | X | X |
| Neurological Exam | X | X |
| 12-Lead ECG | X | X |
| Vital Signs <sup>5</sup> | X | X |
| Hematology, Blood<br>Chemistry, and Urinalysis | X | X |
| Anti-Aducanumab Ab | X | X |
| Coagulation Panel | X X | |
| Brain MRI <sup>6</sup> | X X | |
| C-SSRS-SLV | X X | |
| Concomitant Therapy and Procedures | Monitor and record continuously throughout the study | |
| SAE Reporting | Monitor and record continuously throughout the study | |
| AE Reporting | Monitor and record continuously throughout the study | |

<sup>1</sup>Clinical efficacy assessments (MMSE, CDR, ADAS-Cog13, ADCS-ADL-MCI, NPI-10, RUD-Lite, QoL-AD) have been removed from the Early Termination Visit and safety follow-up visit to reduce participant burden.

<sup>3</sup>If it has been more than 12 weeks since the participant's last dose, participants who had discontinued treatment early but had agreed to remain in the study (following the Table 3 Schedule of Activities in the protocol) should complete this Follow-up visit within 30 days of the clarification letter.

<sup>5</sup>Vital signs will include SBP, DBP, heart rate, body temperature, and respiratory rate. Vital signs will be measured with the participant supine and after the participant has been resting for at least 10 minutes. <sup>6</sup>If an MRI is performed within 14 days of the ET visit, the MRI can be omitted at the ET visit.

#### 2.2.6. Sample Size Considerations

The sample size was mainly based on results from the primary analysis of Study 221AD302. Results from the post-PV4 population (i.e., the 221AD302 and 221AD301 protocol amendment in which the high dose of aducanumab was increased from 6 mg/kg to 10 mg/kg) in pooled data from Studies 221AD302 and 221AD301 were also considered. A total sample size of 1512 participants was planned to have approximately 90% power to detect a mean difference of 0.48 in change from baseline CDR-SB at Week 78 between the 2 treatment groups. This power

<sup>&</sup>lt;sup>2</sup>All participants enrolled in the study are to return to the study site at 12 weeks after the last dose of study treatment for Follow up/End of Study visit. The follow-up visit is important and is intended to monitor the participant after a washout period that is based on the drug's half-life. However, if a study participant with their healthcare provider decides to initiate a disease-modifying Alzheimer's treatment outside of the clinical trial prior to completing all mandated protocol study visits, then the participant should withdraw from the study as per protocol (Protocol Section 8.3, Withdrawal of Participants from Study). For these patients when they are withdrawn, no further study visits should be completed.

<sup>&</sup>lt;sup>4</sup>Pregnancy testing will only be required for women of childbearing potential.

calculation was based on a 2-sided t-test assuming equal variance with a final significance level of 0.05, an SD of 2.33, a dropout rate through Week 78 of 27%, and a randomization ratio of 2:1. The assumed mean difference of 0.48 between the 2 treatment groups represented an approximately 24% reduction in the placebo mean change from baseline at Week 78 if the placebo mean change is estimated to be 2.

In the original study design per protocol, a blinded assessment of the pooled SD for the primary efficacy endpoint may be performed approximately 3 months prior to the completion of enrollment and the sample size may be increased as a result. The sample size could also be increased using internal and external clinical study results that become available after the start of this study. In addition, the sample size may be increased if the dropout rate through Week 78 is estimated to exceed 27%. The sample size will not be reduced based on this assessment.

Following the study early termination decision on 31 January 2024, the blinded assessment of the pooled SD will not be conducted.

#### 3. Definitions

#### 3.1. Dates and Points of Reference

- Study Day 1: the date of the first dose of study treatment (aducanumab or placebo)
- Study Day
  - For a date on or after Study Day 1
     Study Day = (Date of Interest) (Study Day 1) + 1
  - For a date before Study Day 1Study Day = (Date of Interest) (Study Day 1)
- First dose date and last dose date

Unless otherwise specified, the first dose date is equivalent to study Day 1 defined above, the last dose date is the date of the last administration of study treatment.

• End of Treatment (EOT)

EOT date is the last dose date, i.e., Week 104 for treatment completers and at any time during the placebo-controlled (PC) treatment period for early study treatment terminators.

• Early Termination (ET)

Participants who are withdrawn from the study after receiving  $\geq 1$  dose(s) of study treatment should complete the ET visit after the reason for withdrawal is identified. For such participants, efficacy assessments specified at the ET visit are not required if the participant discontinues treatment within 3 months of the previous efficacy assessment visit, and no significant changes in cognitive status are suspected by the Investigator; the site should notify the Sponsor and Medical Monitor in such cases. Participants who are withdrawn from the study are also to return to the site for a FU visit 18 weeks after receiving their last dose of study treatment. Participants should undergo an ET visit unless withdrawal is due to death or withdrawal of consent.

Following the study early termination decision on 31 January 2024, all study participants should complete an ET visit within 30 days after their last dose.

The ET visit date refers to the date of visit for the ET visit.

• End of Study (EOS)

For participants who complete the study, the EOS visit is defined as the Week 122 visit; for participants who early terminate in the study, the EOS visit is defined as the scheduled follow-up (FU) visit, 18 weeks after their final dose.

Following the study early termination decision on 31 January 2024, study participants were required to perform a FU visit 12 weeks after their last dose, instead of 18 weeks.

The EOS date is the End of Study date recorded on the End of Study eCRF page.

• Visit window for analysis

For data that are summarized by visit, assessment from all scheduled visits and unscheduled visits will be mapped to an appropriate analysis visit using a windowing scheme as described in Section 9.1.

## 3.2. Study Treatment

Participants will be assigned to 1 of 2 treatment groups in a 2:1 ratio of aducanumab or placebo administered IV Q4W, respectively. Treatment is initiated via titration, which has been demonstrated to result in a lower incidence of ARIA. Titration will start at 1 mg/kg and will escalate to 3, 6 and 10 mg/kg.

Study treatment in this SAP, unless otherwise specified, refers to the blinded treatment of either aducanumab or placebo that is administrated based on the dosing regimen in this study. Throughout this SAP, study treatment and study drug are equivalent and used interchangeably.

#### 3.3. Study Periods

• Study baseline period

The study baseline period is defined as the period from Screening Visit 1 to the day prior to the first administration of study treatment.

• On treatment period

On treatment period is defined as the period from the first administration of study treatment to 28 days after the last administration of study treatment.

Baseline value

Baseline value is defined as the most recent non-missing measurement collected prior to Study Day 1 dose date/time. If the time of the measurement is missing, measurements taken on Day 1 are considered as prior to Study Day 1 dose for the following data domains: demography, disease history, disease activity and characteristics, clinical endpoint, ECG, laboratory test result, medical history, physical examinations, participant status, and vital signs. Exceptions are specified as below:

- Tau PET baseline value is defined as the most recent non-missing measurement relative to Study Day 1 dose date/time and collected prior to the third dose date or scheduled Week 12 visit date whichever comes first for participants who received more than one dose of study treatment, or within 84 days of the first dose for participants who only received one dose of study treatment, or as the last non-missing measurement collected during screening for not dosed participants.
- Change from baseline is defined as post-baseline value minus baseline value
- Percent change from baseline is defined as post-baseline value minus baseline value then divided by baseline value
- Treatment Emergent

An adverse event is regarded as treatment emergent if the event has onset date/time on or after the first dose date/time of study treatment, or was reported prior to the first

dose and subsequently worsens in severity after first dose date. Additional criteria to determine treatment emergent are described in <u>Section 5.7.1.1</u>.

## 3.4. Key Derived Variables

# 3.4.1. Composite Score Derivation of CDR Subscores and CDR Global Score

The CDR is comprised of 6 domains: Memory, Orientation, Judgment and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care. CDR-SB is the sum of the scores for these 6 domains. In addition, two CDR subscores have been proposed [Tractenberg 2005]: a "cognitive" subscore equaling the sum of the Memory, Orientation, and Judgment and Problem Solving box scores, and a "functional" subscore equaling the sum of Community Affairs, Home and Hobbies and Personal Care box scores.

The CDR global score is a composite score obtained by combining the 6 box scores using a scoring algorithm that weights memory as the primary domain and all other domains as secondary [Morris 1993].

#### 3.5. Stratification Factors

The study randomization stratification factors and corresponding categories are listed as follows:

- Geographical region:
  - o North/South America
  - o Europe/Australia
  - o Asia (Korea/Japan)
  - o China
- Baseline disease stage:
  - o MCI due to Alzheimer's disease
  - o Mild Alzheimer's disease dementia
- ApoE ε4 status:
  - o Carrier
  - o Noncarrier

#### 3.6. Analysis Sets

#### Randomized Set

The randomized set includes all the participants who were randomized.

#### **Full Analysis Set (FAS)**

The FAS includes all participants who were randomized and received at least 1 dose of study treatment (aducanumab or placebo). In analyses performed on the FAS, participants will be analyzed, based on the intention-to-treat principle, according to their randomized treatment assignment regardless of treatment received.

#### Safety Analysis Set

The Safety Analysis Set includes all participants who were randomized and received at least 1 dose of study treatment (aducanumab or placebo), essentially the same set of participants included in the FAS. In analyses performed on the Safety Analysis Set, participants will be analyzed according to their actual treatment received.

#### Safety MRI Analysis Set

The Safety MRI Analysis Set includes all participants who were randomized and received at least 1 dose of study treatment (aducanumab or placebo) and had at least one post-baseline MRI assessment.

# Immunogenicity Analysis Set

The immunogenicity analysis set is defined as all participants in the safety analysis set who had at least 1 postdose sample evaluated for immunogenicity.

#### 4. List of Planned Study Analyses

Below is a list of planned study analyses per protocol.

#### 4.1. Interim Analysis

According to the protocol, interim analyses for superiority may be performed after approximately 60% of the participants have completed the 18-month visit (or discontinued). The alpha level at the interim analysis will be determined using the O'Brien-Fleming boundary approach. The alpha level for the final analysis will be adjusted to achieve an overall type I error of 0.05.

If an interim analysis is performed, the interim analysis will be performed by an independent group external to the Sponsor that will not be involved in the conduct of the study after unblinding. A potential role for the IDMC in this interim analysis will be fully described in the IDMC charter. The aim of this interim analysis is to allow the possibility to verify the clinical treatment benefit of aducanumab early.

If an IA is to be performed, prior to the unblinding for interim analysis, the SAP for the interim analysis will be finalized and signed off. The criteria for determining superiority for the interim analysis will be defined in the interim analysis SAP. This is to ensure that all interim analysis statistical analyses will be pre-specified before the interim analysis.

Following the study early termination decision on 31 January 2024, the optional interim analysis will not be conducted.

#### 4.2. Primary Analysis

The primary analysis (PA) of the study will be conducted when all the participants have had an opportunity to complete the Week 78 visit. After the last patient completes Week 78, the data will be soft locked, and all efficacy endpoints and available safety data will be analyzed while the study is ongoing and continues to capture efficacy, safety, and immunogenicity data beyond Week 78. The PA aims to address all study objectives that use data up to Week 78. This primary analysis will support registration with regulatory agencies. Analyses of Week 78 endpoints will only include data up to Week 78 visit.

This unblinded analysis will be performed by a small internal independent team (separate from the study team).

Following the study early termination decision on 31 January 2024, the planned primary analysis will not be conducted.

#### 4.3. Final Analysis

The final analysis (FA) of the study will be conducted at the end of the study after the last participant completes the last visit of the study and the final database is locked. The FA will evaluate all efficacy endpoints and available safety data, and a review of the complete efficacy and safety collected during the entire study is included.

Following the study early termination decision on 31 January 2024, the final analysis will be conducted at the end of the study after the last participant completes the last visit of the study and the final database is locked following the study conduct that was described in Section 2.2.3. All analyses specified in this SAP will be conducted in the FA with all data collected during the entire study and available in the database.

#### 5. Statistical Methods for Planned Analyses

# 5.1. General Principles

#### 5.1.1. High Level Description of Analyses

This SAP defines the analysis scope for FA. This SAP document supersedes the statistical section in the protocol and provides details for those analyses pre-specified before any planned study unblinding of the Biogen/IQVIA blinded team and before the final database lock. Additional ad hoc analyses may be conducted if needed after data unblinding at the final database lock. If there are any significant modifications in the SAP after data unblinding at the final database lock, those must be documented in the clinical study report accordingly.

Summary tables will be presented using descriptive summary statistics. For continuous endpoints, summary statistics will generally include number of participants with data, mean, standard deviation, median, 25% percentile, 75% percentile, minimum and maximum. For categorical endpoints, this will generally include number of participants randomized or dosed, number with data, and the percent of those with data in each category.

As mentioned in Section 1., due to the early termination of the study, an abbreviated CSR is planned. Accordingly, many endpoints will not be summarized. The data that will be summarized are full safety data, and data on disposition, baseline, demographics, exposure, protocol deviations and CDR-SB. Also, any listings that are routinely produced for Biogen clinical studies will not necessarily be mentioned in this SAP.

There will be no statistical testing for any endpoints.

The statistical software, SAS® version 9.4 or above will be used for all summaries and analyses.

# 5.1.2. Handling of Missing Data on Clinical Measures

If any of the individual items for the CDR-SB, ADAS-Cog13, ADCS-ADL-MCI, and MMSE are missing, the total score of the corresponding endpoint will be imputed by prorating the observed scores [van Ginkel 2010].

For ADAS-Cog 13, if 3 or fewer of 13 items (<25%) are missing, the total score will be imputed by the following algorithm: Total score = total score from the completed items × [maximum total score (=85) / maximum total score for the completed items]. The imputed number will be rounded up to the nearest integer. If more than 3 items are missing, the total score of ADAS-Cog 13 at that visit will be considered missing.

For ADCS-ADL-MCI, if 4 or fewer of 18 items (<25%) are missing, the total score will be imputed by a similar algorithm as that for ADAS-Cog 13. The imputed number will be rounded up to the nearest integer. If more than 4 items are missing, the total score for ADCS-ADL-MCI at that visit will be considered missing.

The same imputation algorithm will be applied to CDR-SB and MMSE: if only 1 box (of 6) of CDR is missing or if only 2 or fewer items (out of 11) are missing for MMSE. If the score from more than 1 box of CDR, or more than 2 items of MMSE is not available, the CDR-SB or MMSE at that visit will be considered missing.

The total score of NPI-10 will be imputed using the same prorating principle if only 1 item (out of 10) is missing.

#### 5.2. Participant Accountability

Disposition of participants will be summarized, and the summary data will include number (%) of participants randomized and dosed, number (%) of participants who completed the treatment/study, number (%) of participants who discontinued treatment and/or withdrew from study. For participants who discontinued treatment and/or withdrew from study, the reasons for discontinuation and/or withdrawal, and days on treatment and days on study will be summarized and listed.

#### 5.3. Demographic and Baseline Characteristics

The demographic data including age, gender, ethnicity, race, region, height, weight, and body mass index (BMI) will be summarized. Age will also be categorized and presented using the following subgroups: <60, 60-70, 71-80, 81-85, >85.

Summary of the baseline characteristics of AD includes laboratory ApoE ε4 status (carrier or non-carrier), baseline clinical stage (MCI due to AD or mild AD), baseline clinical assessment including CDR-SB, CDR cognitive subscore, CDR functional subscore, CDR global score, MMSE, ADAS-Cog 13, ADCS-ADL-MCI, NPI-10, amyloid PET SUVR, tau PET SUVR (available in a subset of sites and participants), number of years of formal education, number of years since first AD symptom, number of years since diagnosis of AD, AD treatment use that was stopped prior to entering the study (yes or no) and AD symptomatic medication use at baseline (yes or no). ApoE ε4 carrier will be further classified as homozygote and heterozygote. MMSE will also be categorized by the following subgroups: <24, 24-26, 27-30.

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The number (%) of participants with history (including both ongoing and not ongoing medical conditions) will be summarized by system organ class and preferred term.

Previous treatment of AD stopped prior to the date of first infusion, duration of previous therapies and reason for stopping treatment will be summarized by treatment group.

The data will be summarized by treatment groups for participants in FAS. Participants listings will be generated for demographics and baseline characteristics.

Note that ApoE ε4 status is defined as follows:

• ApoE ε4 carrier: ε2/ ε4, ε3/ ε4, ε4/ ε4

o Heterozygote:  $\varepsilon 2/\varepsilon 4$ ,  $\varepsilon 3/\varepsilon 4$ 

Homozygote: ε4/ ε4

• ApoE  $\varepsilon$ 4 noncarrier:  $\varepsilon$ 2/ $\varepsilon$ 2,  $\varepsilon$ 2/ $\varepsilon$ 3,  $\varepsilon$ 3/ $\varepsilon$ 3

#### **5.4. Protocol Deviations**

Protocol deviations identified during site monitoring will be captured in a Protocol Deviation log and categorized as major or minor deviations based on Protocol Deviation Classification (see Section 9.2). The major protocol deviations will be summarized for FAS participants by treatment groups. Major protocol deviations for all FAS participants will be listed. Major protocol deviations related to coronavirus disease (COVID-19) may also be summarized and listed.

A listing will be generated for subjects with protocol alternations due to COVID-19, based on the data on the protocol alternations due to COVID-19 collected from the COVID-19 Impact log CRF page.

A listing will be generated for subjects whose treatment assignments were released to the investigators and designated site staff prior to the final database lock, with the date of treatment assignment release presented. See <u>Section 2.2.2.</u> for details about this unblinding procedure.

### 5.5. Study Treatment Exposure and Concomitant Medications

#### 5.5.1. Study Drug Exposure and Study Drug Compliance

A summary table of study drug exposure and compliance will be provided for participants in FAS. Number of infusions (aducanumab or placebo) received will be summarized as a categorical variable (categories of 1-5, 6-10, 11-15, 16-20, 21-26, and >26) as well as a continuous variable. Number of weeks on study treatment (aducanumab or placebo), calculated as (date of last dose – date of first dose +29)/7, will be summarized as a categorical variable (every 8 weeks) as well as a continuous variable. Percentage of study treatment taken up to the last dose, calculated as (the actual number of infusions / by the number of infusions a participant is expected to take until the date of last infusion) ×100, will be summarized as a continuous variable.

Due to the use of a titration regimen in the study and possible dose suspension due to ARIA, another summary table will be provided including the following information in the study: number of infusions at each dose level (1 mg/kg, 3 mg/kg, 6 mg/kg and 10 mg/kg, respectively) summarized as a categorical variable as well as a continuous variable, number of participants with dose increase (placebo to 1 mg/kg, 1 to 3 mg/kg, 3 to 6 mg/kg and 6 to 10 mg/kg, respectively), maximum dose level received, and cumulative dose (as a continuous variable).

A listing of study drug administration records for placebo participants who received any doses of active treatment will be provided.

A listing of subjects whose actual treatment group is different from their randomized treatment group will be provided.

#### 5.5.2. Concomitant Medications

The number (%) of participants taking concomitant medication and non-drug therapies will be summarized for participants in FAS. Concomitant medications and non-drug therapies will be listed.

All concomitant medications will be coded using the World Health Organization (WHO) medication dictionary. All concomitant non-drug therapies will be coded using the MedDRA dictionary. A concomitant medication/therapy will be defined as any therapy that was taken on or after the day of the first dose of study drug. This includes therapies that start prior to the initiation of the first dose if their use continues on or after the date of first dose. To define concomitant use for therapies with missing start or stop dates, the following additional criteria will be used:

- If both the start and stop dates of a therapy are missing, that therapy will be considered concomitant.
- If the start date of a therapy is missing and the stop date of that therapy fall on or after the date of the first dose, that therapy will be considered concomitant.

- If the start date of a therapy is prior to the date of the first dose and the stop date of that therapy is missing and the therapy is listed as ongoing, that therapy will be considered concomitant, or
- If the start date of a therapy is prior to the date of the first dose and the stop date of that therapy is missing and the therapy is not listed as ongoing, that therapy will be considered non-concomitant.

For a therapy with a partial start date, the year/month of the therapy date will be compared to that of the first dosing date to determine whether the therapy is concomitant.

AD symptomatic medications taken concomitantly at baseline are defined as AD symptomatic medications that were being taken at the time of the first dose, i.e., started prior to the first dose and continued until after the first dose. AD symptomatic medications are defined as anticholinesterase (cholinesterase inhibitors) and memantine drugs in the WHO medication dictionary (version: WHODrug Global B3 Sep2023 or a later version if applicable). The number (%) of participants taking concomitant AD symptomatic medications at baseline, number of participants using Cholinesterase inhibitors only, Memantine only, or both at the baseline will be summarized by treatment group for FAS.

# 5.6. Efficacy Endpoints

A summary table of change from baseline by visit in CDR-SB will be presented using descriptive summary statistics, on the FAS.

No statistical modeling will be performed.

## 5.7. Safety Endpoints

#### 5.7.1. Adverse Events

#### **Analysis Methods**

AEs will be analyzed based on safety analysis set. All AEs will be analyzed based on the principle of treatment emergence. A treatment-emergent AE is defined as an AE that started or worsened after the start of the first dose of study treatment.

To define treatment emergence for AEs with missing start or stop date or time the following additional criteria will be used:

- If both the start and stop dates for a particular AE are missing, then that AE is considered treatment emergent;
- If the start date for a particular AE is missing and the stop date/time falls after the first dose date/time, then that AE is considered as treatment emergent;
- If the start date for a particular AE was the same as the first dose date, and the start time was missing, then that event is considered treatment emergent.

For AEs with a partial start date, the year/month of the event date will be compared to that of the first dosing date to determine whether the event is treatment emergent.

In general, AEs will be analyzed based on incidence proportion. The incidence proportion (%) is defined as the number of subjects with an event divided by the total number of subjects in the analysis population. In determining incidence proportion, both single occurrence and multiple

occurrences of events will be counted as one incidence in the numerator. In the remainder of this document and in table titles, incidence proportion may be referred to simply as "incidence".

Adverse events are coded using the MedDRA dictionary. This coding system provides more than five levels to classify AEs. In general, AEs will be presented by SOC and PT but other classifications may be used if warranted.

An overall summary of AEs will be provided by treatment group and by treatment group stratified by ApoE status. This will generally include the following numbers and percentages of subjects: with any AE, with any AE by maximum severity, with any related AE (related to study drug as assessed by the investigator), with SAE, with related SAE (related to study drug as assessed by the investigator), with AE leading to drug discontinuation, with AE leading to study withdrawal, and fatal events.

#### 5.7.1.1. Common Adverse Events

<u>Table 2</u> lists the planned analyses of all AEs, most frequently reported AEs, related AEs (related to study drug as assessed by the investigator), and AEs by severity. All analyses will present incidence proportion by treatment group. Where indicated, the analyses will be repeated by treatment group stratified by ApoE status.

Table 2 Planned Analyses of all AEs, most frequent reported AEs, related AEs, and AEs by severity.

| Analyses of AE incidence proportion | Repeat stratified by ApoE status? |
|---|---|
| AEs by SOC/PT by descending frequency | Yes |
| AEs at least 2% higher in incidence for aducanumab | No |
| compared to placebo by SOC/PT | |
| AEs with an incidence of 5% or more by PT | Yes |
| Severe AEs by SOC/PT | Yes |
| AEs by maximum severity by SOC/PT | Yes |
| Related AEs by SOC/PT | Yes |

A listing presenting all adverse events will be provided containing the following information: participant number, investigator term, PT with reference ID, onset date, onset study day, end date, end study day, duration of AE (in days), outcome, severity, relation (related to study drug as assessed by the investigator), symptom of ARIA (yes/no), serious (yes/no), study withdrawal (yes/no), concomitant treatment (yes/no), and action on study treatment.

A listing of all adverse events related to amyloid PET ligand, related to tau PET ligand or related to lumbar puncture based on data on adverse event CRF page will be provided.

A listing of non-treatment emergent adverse events will be given too.

#### 5.7.1.2. Deaths

Adverse events with fatal outcome will be summarized by SOC/PT, by treatment group and stratified by ApoE status. A listing of deaths will be provided.

#### **5.7.1.3.** Serious Adverse Events

<u>Table 3</u> lists analyses for incidence proportion for SAEs by treatment group. A listing of SAE will also be provided.

Table 3 Analyses of Incidence Proportion for SAE

| Analysis | Repeat stratified by ApoE status? |
|------------------------|-----------------------------------|
| SAEs by SOC/PT | Yes |
| Related SAEs by SOC/PT | Yes |

#### 5.7.1.4. Other Significant Adverse Events

Analysis of other significant AEs will focus on AEs that lead to a substantial intervention, including premature discontinuation of study treatment and withdrawal from study. Adverse events leading to treatment discontinuation will be summarized by SOC/PT, by treatment group and stratified by ApoE status. The same analyses will be repeated for AEs leading to study withdrawal.

Additional summary will be provided for AEs that lead to drug interruption and drug withdrawal.

A separate summary will be provided for ARIA leading to treatment discontinuation as these were protocol-mandated in some circumstances.

Listings of adverse events that led to discontinuation of study drug and adverse events that led to withdrawal from the study will be provided.

# 5.7.1.5. Adverse Events of Special Interest

An AE of special interest is an AE of scientific and medical concern specific to this study, for which ongoing monitoring and reporting is required.

Radiographic ARIA (ARIA-E and ARIA-H), as well as any symptoms of ARIA, are considered AEs of special interest and will be entered on the Adverse Event of Special Interest CRF within 72 hours following the receipt of abnormal MRI findings from the central MRI reader.

In order to guarantee uniformity in ARIA reporting, the AE eCRF has a set verbatim term for cases of ARIA. The verbatim terms together with the corresponding MedDRA preferred terms are shown in Table 4.

Table 4 Verbatim Terms and MedDRA Preferred Terms

| AESI | Verbatim term | MedDRA preferred term |
|--------|------------------------|-----------------------------|
| ARIA-E | Asymptomatic ARIA-E or | Amyloid related imaging |
| | Symptomatic ARIA-E | abnormality-oedema/effusion |

| AESI | Verbatim term | MedDRA preferred term |
|---|---|---|
| ARIA-H | Asymptomatic ARIA-H | Amyloid related imaging |
| microhemorrhage | (Microhemorrhage) or | abnormality-microhaemorrhages and |
| | Symptomatic ARIA-H | haemosiderin deposits |
| | (Microhemorrhage) | _ |
| ARIA-H | Asymptomatic ARIA-H | Superficial siderosis of the central |
| superficial | (Superficial Siderosis) or | nervous system |
| siderosis | Symptomatic ARIA-H (Superficial | |
| | Siderosis) | |
| Cerebral | Cerebral Hemorrhage > 1cm | Cerebral hemorrhages > 1cm refers |
| hemorrhage > | | to Intraparenchymal hemorrhages in |
| 1cm | | the eCRF, and could be coded to |
| | | various preferred terms, depending |
| | | on type of hemorrhage and location |
| | | of hemorrhage. |

Seizures, falls, and hypersensitivity reactions are also considered AEs of special interest.

# 5.7.1.6. ARIA Data Handling Principles

If the radiographic severity of an ARIA event increases or the event changes from asymptomatic to symptomatic, additional AE records will be added to eCRF to capture the change with new start/end AE dates (the end date of the previous record will be the start date of the next record). For analysis, records with changes in severity or symptomatic status are considered as a single ARIA event. The severity/symptomatic status for that event is defined as the worst level among all the AE records that belong to that event.

In general, the start date of the event is the earliest start date among the AE records for the ARIA event, and the end date is the latest end date.

If the same type of ARIA event happens again after the previous event has ended, then it is considered a recurrent event. Recurrent events will be referred to as the second event, the third event, etc.

If the duration based on MRI for an ARIA-E event overlaps with the duration based on MRI for an ARIA-H event, then these two ARIA events will be defined as concurrent.

If a subject experienced ARIA-E but no ARIA-H then this ARIA-E event will be defined as isolated, and similarly for ARIA-H.

The MRI duration of an ARIA event is determined based on MRI assessments. The start date is the date of the MRI assessment that initially identifies the ARIA event, and the end date is the date of the MRI assessment that shows the complete resolution of this ARIA event (in the case of ARIA-E), or ARIA being stable (in the case of ARIA-H). Stable was defined as 'No change' or 'decrease' in number, size, severity, or number of locations of ARIA-H microhemorrhage or ARIA-H superficial siderosis between 2 consecutive MRIs.

The AE eCRF data will be used as the primary source for the ARIA analysis as it contains the complete information of ARIA as well as associated symptoms. The safety MRI data collected

under the 'Neurological Examination' eCRF page will only be used for specific analyses that require information that was not available in the AE eCRF.

## 5.7.1.7. Analysis of Adverse Events of Special Interest

ARIA (ARIA-E, ARIA-H) and cerebral hemorrhage > 1cm events will be summarized based on the Safety MRI Analysis Set. The incidence of ARIA events tables will summarize the number of subjects with any ARIA, ARIA-E, any ARIA-H, ARIA-H microhemorrhage, ARIA-H superficial siderosis, subjects experiencing both ARIA-E and ARIA-H, concurrent ARIA-E and ARIA-H, isolated ARIA-E and isolated ARIA-H.

Cerebral hemorrhage >1 cm will be summarized. Cerebral hemorrhages >1 cm will be identified by the eCRF and by using a customized MedDRA query, consisting of selected preferred terms within the Standardized MedDRA Query (SMQ) of "Haemorrhagic central nervous system vascular conditions (SMQ)" (narrow search). The customized query SMQ list may be modified based on newer version of MedDRA when available and safety team's discretion.

Seizures, hypersensitivity, and fall events will be summarized on the Safety Analysis Set. Seizures will be identified using a customized MedDRA query, consisting of selected preferred terms within the Standardized MedDRA Query (SMQ) of "Convulsions (SMQ)" (narrow search). ARIA status of subjects with seizures will be presented, splitting by the number of subjects with non-evaluable ARIA status (no post-baseline MRI), subjects with no ARIA event during the study and subjects who experienced ARIA during the study.

Hypersensitivity events will be identified using a customized MedDRA query, consisting of selected preferred terms within the Standardized MedDRA Query (SMQ) of "Hypersensitivity (SMQ)" (narrow scope). The hypersensitivity SMQ list may change due to newer version of MedDRA and at safety team's discretion.

Falls will be identified based on the preferred term "Fall" and number of falls will be presented by treatment group.

Other analyses of AEs within this SMQ may be performed, including exploration of potential association with ARIA-E. Analyses to describe and characterize the incidence of AESIs are listed in Table 5 below. Unless otherwise specified, results will be presented by treatment group.

Table 5 Analyses to Describe Incidence of AESIs and to Characterize AESI Events

| Analysis |
|---|
| Incidence of ARIA events |
| Incidence of ARIA events by ApoE e4 genotype |
| Maximum MRI severity and worst symptomatic status of ARIA events |
| Maximum MRI severity and worst symptomatic status of ARIA events by ApoE genotype |
| Maximum MRI severity and worst symptomatic status of ARIA events among participants with |
| ARIA |
| Onset of ARIA events |
| Resolution of ARIA-E and stabilization of ARIA-H |
| Recurrent ARIA-E |
| ARIA-related adverse events by SOC/PT |

| <b>A</b> | - | • |
|----------|-----|------|
| An | alv | ysis |

Summary of symptomatic ARIA

Summary of serious and severe ARIA and symptoms

Serious or severe ARIA-related adverse events by PT

Cerebral hemorrhage > 1cm

Haemorrhagic CNS vascular conditions events by PT<sup>12</sup>

Haemorrhagic CNS vascular conditions events excluding subdural hematomas by PT<sup>12</sup>

Hypersensitivity events by PT<sup>13</sup>

Serious hypersensitivity events by PT<sup>13</sup>

Related hypersensitivity events by PT<sup>13</sup>

Seizures by PT<sup>13</sup>

Falls<sup>13</sup>

The following listings will also be provided with the relevant information:

- Listing of MRI assessments for subjects with ARIA-E
- Listing of MRI assessments for subjects with ARIA-H microhemorrhage
- Listing of MRI assessments for subjects with ARIA-H superficial siderosis
- Listing of MRI assessments for subjects with Cerebral hemorrhage > 1cm
- Listing of MRI assessments for subjects with other postbaseline MRI abnormalities
- Listing of MRI assessments for subjects with postbaseline MRI ischemic abnormalities
- Listing of ARIA-related adverse events for subjects with symptomatic ARIA based on Adverse Event CRF
- Listing of haemorrhagic CNS vascular conditions
- Listing of hypersensitivity adverse events
- Listing of seizures
- Listing of falls

#### 5.7.2. Clinical Laboratory Evaluations

Clinical laboratory evaluations include hematology, blood chemistry and urinalysis. Baseline for laboratory parameters is defined as the last available value prior to the first dose.

For each laboratory category, the following analyses will be presented:

- Summaries of actual values by visit and respective figures displaying the mean values by visit
- Summaries of change from baseline by visit
- Summaries of percent change from baseline by visit

<sup>&</sup>lt;sup>1</sup>On safety population.

<sup>&</sup>lt;sup>2</sup>Haemorrhagic CNS vascular conditions event is defined by haemorrhagic central nervous system vascular conditions SMQ (broad and narrow scope).

<sup>&</sup>lt;sup>3</sup>Hypersensitivity reaction event is defined by hypersensitivity SMQ (narrow and broad scope), angioedema SMQ (narrow and broad scope) and anaphylactic reaction SMQ (narrow and broad scope).

<sup>&</sup>lt;sup>4</sup>Seizures event is defined by Convulsions SMQ (broad and narrow scope).

<sup>&</sup>lt;sup>5</sup>Fall event is defined by the preferred Term "Fall".

- Shift from baseline
- Potentially serious hepatotoxicity evaluation will be presented in a figure with respective listing. For subjects with potential serious hepatotoxicity, values over time will also be presented in a figure.

Note: Potentially serious hepatotoxicity is defined as ALT or AST > 3x ULN and total bilirubin > 2x ULN at any time post-baseline, not necessarily concurrent.

Potentially Clinically Significant laboratory abnormalities analyses

For hematology, blood chemistry and urinalysis, the number of subjects with potentially clinically significant laboratory abnormalities post-baseline will be summarized for the parameters provided in Table 6. Subjects need to have at least one post-baseline evaluation and a baseline value not potentially clinically significant (including missing) to be included in the analysis.

Table 6 Criteria to Determine Potentially Clinically Significant (PCS) Laboratory Abnormalities

| Clinical Laboratory Abnormality Criteria | | |
|---|---|---|
| Parameter name | PCS Low | PCS High |
| HEMATOLOGY | | |
| White blood cells | <3.0 x 109/L | >16 x 109/L |
| Lymphocytes | <0.8 x 109/L | >12 x 109/L |
| Neutrophils | <1.5 x 109/L | >13.5 x 109/L |
| Monocytes | N/A | >2.5 x 109/L |
| Eosinophils | N/A | >1.6 x 109/L |
| Basophils | N/A | >1.6 x 109/L |
| Red blood cells | ≤3.5 x 1012/L | ≥6.4 x 1012/L |
| Hemoglobin - Females | ≤95 g/L | ≥175 g/L |
| Hemoglobin - Males | ≤115 g/L | ≥190 g/L |
| Hematocrit - Females | ≤32% | ≥54% |
| Hematocrit - Males | ≤37% | ≥60% |
| Platelet count | ≤75 x 109/L | ≥700 x 109/L |
| BLOOD CHEMISTRY | | |
| Alanine aminotransferase (ALT) | N/A | >3 x ULN |
| Aspartate aminotransferase (AST) | N/A | >3 x ULN |
| Alkaline phosphatase (ALP) | N/A | >3 x ULN |
| Total bilirubin | N/A | >1.5 x ULN |
| Blood urea nitrogen (BUN) | N/A | ≥10.7 mmol/L |
| Creatinine | N/A | ≥176.8 umol/L |
| Sodium | ≤126 mmol/L | ≥156 mmol/L |
| Potassium | ≤3 mmol/L | ≥6 mmol/L |
| Chloride | ≤90 mmol/L | ≥118 mmol/L |
| Bicarbonate | ≤16 mmol/L | ≥35 mmol/L |

| Glucose | ≤2.2 mmol/L | ≥9.7 mmol/L |
|-----------------------------|-------------|-------------|
| Calcium | ≤2 mmol/L | ≥3 mmol/L |
| Phosphorus | ≤0.6 mmol/L | ≥1.7 mmol/L |
| Albumin | ≤25 g/L | ≥625 g/L |
| Total protein | ≤45 g/L | ≥100 g/L |
| <u>URINALYSIS</u> | | |
| Glucose | N/A | ≥++++ |
| Ketones | N/A | ≥++++ |
| Protein | N/A | ≥++ |
| ULN = upper limit of normal | | |

#### 5.7.3. Vital Signs

Vital sign parameters include body temperature, systolic blood pressure, diastolic blood pressure, heart rate, respiration rate, and body weight. Baseline is defined in a similar way as with clinical laboratory parameters.

Clinically relevant post-baseline abnormalities in vital signs will be presented with criteria defined below:

- $< 36 \, ^{\circ}\text{C}$  and  $> 38 \, ^{\circ}\text{C}$  for body temperature
- < 60 bpm and > 100 bpm for pulse
- < 90 mmHg, > 140 mmHg and > 160 mmHg for systolic blood pressure
- < 50 mmHg, > 90 mmHg and > 100 mmHg for diastolic blood pressure
- $\geq$  7% increase and  $\geq$  7% decrease from baseline in weight
- < 12 breaths/min and > 20 breaths/min for respiratory rate

#### 5.7.4. Physical Examination and Neurological Examination

Clinically significant abnormalities found at a physical examination or neurological examination will be reported as AEs and will be included in the analyses of AEs.

#### 5.7.5. Electrocardiograms

The 12-lead electrocardiograms (ECG) data will be summarized using shift table based on subjects with at least one post-baseline ECG assessment and whose baseline ECG assessment was not abnormal. This includes shift from normal or unknown at baseline to abnormal post-baseline, shift from normal or unknown at baseline to not adverse event or abnormal post-baseline, and shift from normal or unknown at baseline to adverse event post-baseline.

The number and percentage of subjects with shifts to abnormal ECG, not adverse events, and subjects with shift to abnormal ECG, adverse events at any time during post-baseline will be summarized. The ECG outlier in the uncorrected QT and Fridericia's corrected QTc intervals are the values exceeding a threshold of particular concern in clinical trials and are defined using criteria listed in FDA guidance - E14 Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs. The number and percentage of subjects

with ECG outlier in the uncorrected QT and Fridericia's corrected QTc interval will be summarized by treatment group.

- Absolute QTc interval prolongation:
  - $\circ$  OTc interval > 450
  - o QTc interval > 480
  - o QTc interval > 500
- Change from baseline in QTc interval:
  - O QTc interval increases from baseline > 30
  - O QTc interval increases from baseline > 60

Baseline is defined in a similar way as with clinical laboratory data. The worst post-baseline value of each subject will be used.

# 5.7.6. Immunogenicity

# 5.7.6.1. Background

#### Definition of baseline value

Baseline value is defined as the latest immunogenicity data collected prior to the first dose. If no immunogenicity data are collected prior to the first dose, baseline value will be treated as antidrug antibody (ADA) negative for immunogenicity analyses.

A summary of treatment-emergent anti-aducanumab positive responses will also be presented using the following definitions:

Post-baseline positive anti-aducanumab antibody responses are defined as treatment-emergent if a subject is either (1) antibody negative at baseline; or (2) antibody positive at baseline but the post-baseline antibody response is more than 2-fold increase in titer compared to the baseline response.

Persistent and transient positive responses for the placebo-controlled period:

Subjects with treatment-emergent positive anti-aducanumab antibody responses in the placebocontrolled period will be further classified as transient positive under the following conditions:

- if only a single positive evaluation occurs which is not at the last available time point
- or if more than 1 positive evaluation occurs < 112 days (16 weeks) apart and there is at least 1 evaluation occurs thereafter;

Subjects with treatment-emergent positive anti-aducanumab antibody responses in the placebocontrolled period will be further classified as persistent positive under the following conditions:

- if more than one consecutive positive evaluation occurs  $\geq 112$  days (16 weeks) apart
- or if a single positive evaluation occurs at the last available time point with no further negative results available

#### 5.7.6.2. Immunogenicity analysis

Immunogenicity analysis set will be used for immunogenicity analysis. Tables will be presented by treatment group. Listings will be presented by treatment group stratified by ApoE status.

A summary table will be presented showing the number of subjects with treatment-emergent anti-aducanumab antibody positive response at any time post-baseline, the number of subjects with treatment-emergent anti-aducanumab antibody positive response at each visit, the number of subjects with persistent and transient response, the number of subjects positive at baseline with a treatment-emergent response and without a treatment-emergent response, and the number of subjects positive post-baseline or at baseline (with or without a treatment-emergent response). A listing of immunogenicity assessments as well as a listing of adverse events for subjects with any anti-aducanumab antibody positive results will also be provided.

#### 5.7.7. C-SSRS

The Columbia Suicide Severity Rating Scale (C-SSRS) is an assessment that evaluates suicidal ideation and behavior.

A summary of post-baseline C-SSRS results will be presented showing:

- The number of subjects with at least one post-baseline C-SSRS assessment
- The number of subjects with suicidal ideation
- Number of subjects with suicidal behavior
- Number of subjects with suicidal ideation or behavior
- Non-suicidal self-injurious behavior

The listing of subjects with post-baseline suicidal ideation, suicidal behavior, or non-suicidal self-injurious behavior, the listing of subjects with post-baseline suicidal ideation, and the listing of subjects with post-baseline suicidal behavior will also be presented.

### 6. Changes from Protocol-Specified Analyses

On 31 January 2024, the early termination of Study 221AD305 was announced. Consequently, protocol-specified final analysis that was designed to verify the clinical benefit of aducanumab will not be performed; only the analyses described in Section 5 will be performed. All protocol pre-specified analysis that were designed to assess the safety of monthly doses of aducanumab will be performed. Specifically, the changes in the planned analysis are as follows:

# 6.1. Primary Endpoint, Key Secondary Endpoints and Secondary Endpoints

Primary endpoint CDR-SB will be summarized. There will be no statistical testing.

The protocol-specified key secondary endpoints and secondary endpoints will not be analyzed.

## 6.2. Tertiary Endpoints

Protocol specified tertiary endpoints individual items of the RUD-Lite and QoL-AD scores will not be analyzed.

Protocol specified tertiary endpoints serum concentrations and PK parameters of aducanumab over time will not be analyzed.
# 7. Summary of Changes from the Previous Version of the SAP

This section is not applicable as there is no previous version of the SAP.

## 8. References

221AD305 ENVISION Clarification Letter 16FEB2024 Final Signed

221AD305 Unblinding Plan v3.4 29APR2024

Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993;43(11):2412–2414.

Tractenberg RE, Weiner MF, Cummings JL, Patterson MB, Thal LJ. Independence of changes in behavior from cognition and function in community-dwelling persons with Alzheimer's disease: a factor analytic approach. Journal of Neuropsychiatry and Clinical Neuroscience. 2005;17(1):51–60.

van Ginkel JR, SijtsmaK, van der Ark LA, & Vermunt, JK. Incidence of missing item scores in personality measurement, and simple item-score imputation. Methodology: European Journal of Research Methods for the Behavioral and Social Sciences, 2010; 6(1), 17-30.

## 9. Appendix

## 9.1. Visit Window

For analyses summarized by visit, data collected during all scheduled and unscheduled visits will be mapped to an appropriate analysis visit using the windowing scheme shown below. If there are 2 or more assessments available in the same analysis window for a participant, the assessment that is closest to the target visit day will be used for analysis. If there are 2 or more assessments in the same analysis window with the same distance from the target visit day, the later assessment will be used.

As illustrated in Section 2.2.2., there are changes in the timing and the assessments to be collected for the safety follow-up visit following the study early termination. Because of these changes, the visit window mapping will vary depending on whether the corresponding assessment is collected at the follow-up visit and if the participant has achieved Week 122 as of January 31, 2024. Specifically:

- (1) If an assessment is not collected in the revised safety follow-up visit, the visit window mapping is not impacted and will be the same for all participants
- (2) If an assessment is collected in the revised safety follow-up visit
  - a. For those participants who have reached Week 122 as of January 31, 2024, the visit window mapping will use the windowing scheme that assumes safety follow-up visit is at Week 122 (18 weeks after Week 104)

    Because Study 221AD305's first participant was randomized and dosed on July 27, 2022, the expected Week 122 visit would have occurred in November 2024. Therefore, as of January 31, 2024, there should be no participants who had Week 122 visit.
  - b. For those participants who have not reached Week 122 as of January 31, 2024, the visit window mapping will use the windowing scheme that the safety follow-up visit is Week 116 (12 weeks after Week 104).

## 9.1.1. Visit Windows for Mapping Efficacy Endpoint CDR-SB

For CDR-SB summaries by visit, data collected during all scheduled and unscheduled visits will be mapped to an appropriate analysis visit using the windowing scheme shown in <u>Table 7</u>. If there are 2 or more assessments available in the same analysis window for a participant, the assessment that is closest to the target visit day will be used for analysis. If there are 2 or more assessments in the same analysis window with the same distance from the target visit day, the later assessment will be used.

Table 6 Visit Windows for Efficacy Endpoint CDR-SB

| Endpoints | Analysis Visit | Target Visit Day | Analysis Visit |
|---|---|---|---|
| | | | Window |
| | Clinical F | Efficacy Endpoint | |
| CDR-SB score | Baseline | 1 | Most recent non-<br>missing pre-dose<br>value |
| | Week 26 | 183 | [92, 266] |
| | Week 50 | 351 | [267, 448] |
| | Week 78 | 547 | [449, 644] |
| | Week 106 | 743 | [645, 798] |
| | Week 122 <sup>1</sup> | 855 | ≥ 799 |

<sup>1:</sup> CDR has been removed from the revised schedule of activities of follow-up visit. Therefore, visit window mapping is not impacted by the revised schedule of follow-up visit.

# 9.1.2. Visit Windows for Mapping Laboratory Parameters

Table 7 Visit Windows for Laboratory Parameters

| Endpoints | Analysis Visit | Target Visit Day | Analysis Visit<br>Window |
|---|---|---|---|
| For participants who h | ave reached Week 122 as | s of January 31, 2024 | |
| Hematology, Blood | Baseline | 1 | Most recent non- |
| Chemistry, and | | | missing pre-dose |
| Urinalysis | | | value |
| | Week 52 | 365 | [2, 546] |
| | Week 104 | 729 | [547, 791] |
| | Week 122 | 855 | ≥ 792 |
| For participants who h | ave not reached Week 12 | 22 as of January 31, 2024 | 1 |
| Hematology, Blood | Baseline | 1 | Most recent non- |
| Chemistry, and | | | missing pre-dose |
| Urinalysis | | | value |
| | Week 52 | 365 | [2, 546] |
| | Week 104 | 729 | [547, 770] |
| | Week 116 | 813 | ≥ 771 |

# 9.1.3. Visit Windows for Mapping Vital Sign Parameters

Table 8 Visit Windows for Vital Sign Parameters

| Endpoints | Analysis Visit | Target Visit Day | Analysis Visit |
|---|---|---|---|
| | | | Window |
| For participants who have reached Week 122 as of January 31, 2024 | | | |
| Vital Signs | Baseline | 1 | Most recent non-<br>missing pre-dose<br>value |
| | Week 4 | 29 | [2, 42] |

| | | T | T-12 -22 |
|---------------------|-----------------------|---------|------------------|
| | Week 8 | 57 | [43, 70] |
| | Week 12 | 85 | [71, 98] |
| | Week 16 | 113 | [99, 126] |
| | Week 20 | 141 | [127, 154] |
| | Week 24 | 169 | [155, 182] |
| | Week 28 | 197 | [183, 210] |
| | Week 32 | 225 | [211, 238] |
| | Week 36 | 253 | [239, 266] |
| | Week 40 | 281 | [267, 294] |
| | Week 44 | 309 | [295, 322] |
| | Week 48 | 337 | [323, 350] |
| | Week 52 | 365 | [351, 378] |
| | Week 56 | 393 | [379, 406] |
| | Week 60 | 421 | [407, 434] |
| | Week 64 | 449 | [435, 462] |
| | Week 68 | 477 | [463, 490] |
| | Week 72 | 505 | [491, 518] |
| | Week 76 | 533 | [519, 539] |
| | Week 78 | 547 | [540, 553] |
| | Week 80 | 561 | [554, 574] |
| | Week 84 | 589 | [575, 602] |
| | Week 88 | 617 | [603, 630] |
| | Week 92 | 645 | [631, 658] |
| | Week 96 | 673 | [659, 686] |
| | Week 100 | 701 | [687, 714] |
| | Week 104 | 729 | [715, 791] |
| | Week 122 | 855 | ≥ 792 |
| For participants wh | o have not reached We | | • |
| Vital Signs | Baseline | 1 | Most recent non- |
| | | | missing pre-dose |
| | | | value |
| | Week 4 | 29 | [2, 42] |
| | Week 8 | 57 | [43, 70] |
| | Week 12 | 85 | [71, 98] |
| | Week 16 | 113 | [99, 126] |
| | Week 20 | 141 | [127, 154] |
| | Week 24 | 169 | [155, 182] |
| | Week 28 | 197 | [183, 210] |
| | Week 32 | 225 | [211, 238] |
| | Week 36 | 253 | [239, 266] |
| | Week 40 | 281 | [267, 294] |
| | Week 44 | 309 | [295, 322] |
| | Week 48 | 337 | [323, 350] |
| | Week 52 | 365 | [351, 378] |
| | Week 56 | 393 | [379, 406] |
| | 11 COR 50 | 1 5 7 5 | [ [272, 100] |

| Week 60 | 421 | [407, 434] |
|----------|-----|------------|
| Week 64 | 449 | [435, 462] |
| Week 68 | 477 | [463, 490] |
| Week 72 | 505 | [491, 518] |
| Week 76 | 533 | [519, 539] |
| Week 78 | 547 | [540, 553] |
| Week 80 | 561 | [554, 574] |
| Week 84 | 589 | [575, 602] |
| Week 88 | 617 | [603, 630] |
| Week 92 | 645 | [631, 658] |
| Week 96 | 673 | [659, 686] |
| Week 100 | 701 | [687, 714] |
| Week 104 | 729 | [715, 770] |
| Week 116 | 813 | ≥ 771 |

# 9.1.4. Visit Windows for Mapping Immunogenicity

Table 9 Visit Windows for Immunogenicity

| Endpoints | Analysis Visit | Target Visit Day | Analysis Visit<br>Window |
|---|---|---|---|
| For participants who ha | ave reached Week 122 a | s of January 31, 2024 | |
| Anti-Aducanumab<br>Ab | Baseline | 1 | Most recent non-<br>missing pre-dose<br>value |
| | Week 12 | 85 | [2, 126] |
| | Week 24 | 169 | [127, 266] |
| | Week 52 | 365 | [267, 455] |
| | Week 78 | 547 | [456, 637] |
| | Week 104 | 729 | [638, 791] |
| | Week 122 | 855 | ≥ 792 |
| For participants who h | ave not reached Week 12 | 22 as of January 31, 2024 | 1 |
| Anti-Aducanumab<br>Ab | Baseline | 1 | Most recent non-<br>missing pre-dose<br>value |
| | Week 12 | 85 | [2, 126] |
| | Week 24 | 169 | [127, 266] |
| | Week 52 | 365 | [267, 455] |
| | Week 78 | 547 | [456, 637] |
| | Week 104 | 729 | [638, 770] |
| | Week 116 | 813 | ≥ 771 |

# 9.1.5. Visit Windows for Mapping Brain MRI

**Table 10** Visit Window for Brain MRI

| Endpoints | Analysis Visit | Target Visit Day | Analysis Visit<br>Window |
|---|---|---|---|
| For participants who h | nave reached Week 122 | as of January 31,2024 | |
| Brain MRI assessment | Baseline | 1 | Most recent non-<br>missing pre-dose<br>value |
| | Week 14 | 99 | [2, 126] |
| | Week 22 | 155 | [127, 182] |
| | Week 30 | 211 | [183, 252] |
| | Week 42 | 295 | [253, 518] |
| | Week 106 | 743 | [519, 798] |
| | Week 122 | 855 | >=799 |
| For participants who h | nave not reached Week | 122 as of January 31, 202 | 24 |
| Brain MRI assessment | Baseline | 1 | Most recent non-<br>missing pre-dose<br>value |
| | Week 14 | 99 | [2, 126] |
| | Week 22 | 155 | [127, 182] |
| | Week 30 | 211 | [183, 252] |
| | Week 42 | 295 | [253, 518] |
| | Week 106 | 743 | [519, 777] |
| | Week 116 | 813 | >=778 |

# 9.2. Protocol Deviation Classification

**Table 11 Summary of Protocol Deviation Classification** 

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| IP administration | IP administered < 21 days from previous dose | Major |
| Concomitant<br>Medications | Change in AD medications during course of the study without completion of the unscheduled AD medication visit before the change or within 30 days after the change (if the investigator is notified after the change already occurs) | Minor |
| Concomitant<br>Medications | The subject used prohibited concomitant medication (or therapies) | Major |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| Randomization | Mis-stratification due to entry error related to disease stage or ApoE carrier status in IRT | Major |
| IP administration | ARIA Dosing Rules not followed as per protocol: includes dose suspended when it should have been continued, dose continued when it should have been suspended, titration schedule not followed upon dose resumption | Major |
| | As this may be noted by the blinded team on infusion notes and/or the unblinded team on the IP preparation documents both may report. This type of PD will need to be reconciled regularly to prevent duplication in the final log and to make sure none are missed. | |
| Laboratory assessment | Required lab samples not done at first ARIA management visit (for each new ARIA) | Minor |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | Follow up phone call / visit not done at unscheduled ARIA visit | Minor |
| Informed Consent and Process | Care partner did not sign consent prior to study participant beginning study procedures. | Major |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | Missed CSF sample at timepoints for CSF substudy participants. | Minor |
| Concomitant<br>Medications | Administration of any disallowed concomitant therapy <u>or</u> non-adherence to the limits of those medications that are permitted but have limitations on use (protocol section 7.7.1.2.1) | Major |
| IP preparation | Mis-dose (underdose) due to rounding errors (not following DHA) or errors in weight calculations | Minor if isolated;<br>Major if there is a<br>trend |
| Exclusion criteria | Exclusionary lab value results but subject was randomized and dosed. | Major Possibly critical depending on whether there is an immediate safety concern from the lab value |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| Inclusion Criteria<br>or Exclusion<br>Criteria<br>(depending on<br>criterion) | Any eligibility assessment other than Inclusion criterion #2, #5, #7 not performed such that eligibility could not be confirmed at the time of enrollment but when done after the fact the participant is confirmed as eligible. NOTE: If participant is confirmed as ineligible follow the classification for ineligible participant | Minor |
| Exclusion criteria | and PD is major. Any confirmed deviation from exclusion criteria such that participant was not eligible for participation. SM is to note which criterion was | Major |
| | violated in the PD text. Note: this does NOT include cases where participants met the exception criteria for malignancy and are eligible for the study following TMA review. | |
| Inclusion Criteria | Any confirmed deviation from inclusion criteria such that participant was not eligible for participation. SM is to note which criterion was violated in the PD text. | Major |
| Inclusion Criteria | Subject not eligible based on scores of CDR,<br>MMSE, RBANS-DMI, as defined by inclusion<br>criterion # 7 | Major |
| Inclusion Criteria | CDR, MMSE, RBANS-DMI not done prior to randomization such that eligibility could not be assessed. | Major |
| Inclusion Criteria | Amyloid PET or CSF not done prior to randomization such that eligibility could not be assessed but participant is confirmed as eligible after the fact. | Major |
| Efficacy | Inconsistent rater used for primary, secondary endpoints if for reasons other than allowed by the protocol | Major |
| Informed Consent and Process | ICF obtained by subject is not in a language understandable by the participant/LAR | Major/ Potentially<br>Critical |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| Informed Consent | Incompat completion of ICE (i.e. subject/core | Minor |
| and Process | Incorrect completion of ICF (i.e., subject/care | IVIIIIOI |
| and Process | partner/LAR/person obtaining consent did not | |
| | provide date of signature; subject/care | |
| | partner/LAR/person obtaining consent noted | |
| | incorrect date of signature; subject/care | |
| | partner/LAR/person obtaining consent printed | |
| | name when should have signed, subject/care | |
| | partner/LAR/person obtaining consent signed on | |
| | line for printed name, printed name on line for | |
| | signature, etc.) | |
| Informed Consent | Subject/informant/legally authorized | Major |
| and Process | representative OR PI/site staff administering | |
| | consent did not sign consent (main or sub study | |
| | prior to procedures covered by that consent being | |
| | performed | |
| Informed Consent | Incorrect or outdated version of ICF signed | Major |
| and Process | (applies to main, sub studies/optional consents and | 1,14,01 |
| | care partner). | |
| IP administration | Site used IP without waiting for confirmation that | Minor or Major (see |
| | it was usable following a temperature excursion | comments) |
| IP administration | Use of IP that was rejected following a | Major |
| ir adillilistration | | Major |
| ID 1 ' ' ' ' | temperature excursion | 3.6 ' |
| IP administration | Titration schedule not respected when preparing IP | Major |
| IP administration | Use of expired IP | Minor |
| Subject IP | Unblinded pharmacist not maintaining appropriate | Major |
| compliance | packaging or labels to allow the UB SM to verify | |
| | IP accountability. | |
| Blinding | IP is not stored in blinded manner or according to | Major |
| | the site's signed Blind Maintenance Plan | |
| | NOTE 10 | |
| | NOTE: if anyone at the site or sponsor/IQVIA | |
| | team has been unblinded as a result of the storage | |
| | issue, follow the PD guidance for treatment | |
| | unblinding | |
| IP conditions | IP storage temperature out of range (2-8 °C). | Minor unless trend |
| IP conditions | Temperature excursions not reported as per | Major |
| | Biogen's process | |
| IP conditions | IP temperature monitoring documentation is not | Minor unless trend |
| | being maintained | |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| Laboratory assessment | Samples not received at the central laboratory according to shipment requirements (frozen samples received ambient; ambient samples received frozen) | Minor |
| Laboratory assessment | Laboratory result not acknowledged by PI, or medically qualified and delegated study personnel in a timely manner. | Minor (unless trending) |
| | NOTE: If delayed lab review potentially impacted eligibility, please refer to the inclusion/exclusion PD guidance. | |
| Laboratory assessment | Pre-dose and/or post-dose PK samples not collected, or not collected within protocol specified time. | Minor |
| Laboratory assessment | Lab specimens temperature log (freezer) is not being maintained nor checked by applicable study personnel. | Minor |
| Laboratory assessment | Coagulation tests not completed per protocol prior to lumbar puncture (within 35 days normally and within 7 days for participants with elevated risk for bleeding) | Major |
| Laboratory assessment | Lab samples not drawn, drawn out of window, or results unavailable | Minor |
| Laboratory assessment | Use of incorrect lab kit. | Minor |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | Participant is eligible per malignancy exceptions noted in the protocol but the SAF was submitted for review retrospectively. | Minor |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | Baseline tau PET scan not done for participant at a mandatory tau site | Minor |
| Exclusion criteria | Participant has been randomized and received first dose of study medication but used allowed chronic concomitant medications at doses that were not been stable for at least 4 weeks prior to Screening Visit 1 and during Screening up to Day 1, or used Alzheimer's disease medications at doses that were not stable for at least 8 weeks prior to Screening 1 up to Day 1 or used allowed chronic | Major |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| 3 1 | concomitant medications that affect cognition at doses that were not stable for at least 8 weeks prior to screening Visit 1 and during screening up to Day 1. | |
| Randomization | Subject enrolled (for treatment) in IXRS but not treated | Major |
| Randomization | Subject randomized to wrong arm due to mis-entry of ApoE ε4 carrier status. | Major |
| IP administration | Wrong study drug dispensed | Major |
| IP administration | Subject received IP despite meeting discontinuation or withdrawal criteria | Major |
| IP administration | Missed infusion not due to ARIA | Major |
| Efficacy | CDR, ADCS-ADL-MCI, ADAS-Cog 13, MMSE, NPI-10 not administered SM may record one PD at the visit level, including all the assessments, as long as there is no difference in the category or severity. A second PD should be included for minor assessments missed at the same visit. | Major |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | Any individual procedure not conducted per protocol requirements (either skipped or out of window) except those noted in the note. SM may record one PD at the visit level, including all the assessments, as long as there is no difference in the category or severity. NOTE: Does not apply to MRI, Infusions, CDR, ADCS-ADL-MCI, ADAS-Cog 13, MMSE, NPI-10, C-SSRS and labs, which, if missed, are considered major PD per this classification document | Minor |
| Safety | Participant dosed based on local read of MRI rather than central read as required by protocol | Major |
| Safety | MRI visit or individual MRI not done (scheduled or unscheduled ARIA visit) | Major / potentially critical |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| Safety | MRI conducted on subsequent participants without receiving passing QC report on first in-vivo scan | Major |
| Safety | Infusion conducted prior to receipt and/or review of MRI central read results or QC report | Major / potentially critical |
| Efficacy | Assessment performed by non-qualified rater (this applies to all scales for which MedAvante is confirming qualification and not only cognitive scales | Major |
| Efficacy | CDR, ADCS-ADL-MCI, ADAS-Cog 13, MMSE, NPI-10 administered out of window (OOW) SM may record one PD at the visit level, including all the assessments, as long as there is no difference in the category or severity. A second PD should be included for minor assessments missed at the same visit. | Minor |
| IP preparation | Overdose of study medication, includes mis-dose (overdose) due to rounding errors or errors related to weight calculation | Major |
| IP administration | Overdose Form not submitted to IQVIA Lifecycle Safety within 24 hours of site being made aware of an overdose. | Major |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | PET scan conducted on subsequent participants without receiving passing QC report on first invivo scan | Minor |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | Missed PET scan at timepoints for PET substudy participants. | Minor |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | Ligand dose administration error for either PET | Major |
| Safety | Pregnancies not appropriately reported within 24 hours of study site staff becoming aware of the pregnancy. | Major |
| Efficacy | Administration of rating scales over the telephone. | Major |
| Efficacy | CDR raters were performing other assessments on subjects they performed CDRs for. | Major |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| Efficacy | Independent Rater 2 performed CDR on participant for which they already performed ADAS-Cog, ADCS-ADL-MCI, MMSE, RBANS, C-SSRS | Major |
| Efficacy | Independent Rater 2 performed CDR on participant for which they already performed NPI, EQ-5D-5L, Rud-Lite, QoL-AD | Minor |
| Efficacy | RDV / DSF rater performed RBANS or C-SSRS on the same subject (PV2) | Minor |
| Efficacy | RDV / DSF rater performed CDR, ADAS-Cog 13, ADCS-ADL-MCI, MMSE, NPI, EQ-5D-5L, Rud-Lite, QoL-AD on the same subject | Major |
| Safety | C-SSRS not administered or administered out of window (applies to both protocol scheduled and ARIA unscheduled visits) | Major |
| Informed Consent and Process | Participant not reconsented in a timely manner, expected at the first clinical visit following availability of a newly EC/IRB approved ICF (applies to main, sub study and optional ICFs) | Major |
| Informed Consent and Process | Care partner is not reconsented in a timely manner, expected at the first care partner visit following receipt of a newly EC/IRB approved care partner ICF. | Minor |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | Re-screening not approved in advance by Medical | Major |
| Study assessments criteria | Essential baseline evaluations were not performed prior to initiation of study drug. CDR-SB ADCS-ADL-MCI ADAS-Cog13 MMSE NPI-10 | Major |
| Study assessments criteria | Dose reduction or dose increase administered by PI/sub-I when protocol requires return to same dose that participant was given prior to the ARIA event following temporary discontinuation of IP following ARIA event | Major |
| Study assessments criteria | Primary endpoint assessment CDR-SB not conducted or administered at a study visit, as per protocol. Please note that deviation will not apply for any cognitive assessments that were not | Major |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| | administered or completed, due to subject's decline in cognition. | |
| Study assessments criteria | Secondary endpoint assessments PET scan not conducted or administered at a study visit, as per protocol. Please note that deviation will not apply for any cognitive assessments that were not administered or completed, due to subject's decline in cognition. | Major |
| Study assessments criteria | ARIA management not being followed as per protocol specifications. | Major |
| Study assessments criteria | Study MRIs missed. | Major |
| Safety | SAEs or AESI (ARIA, Fall, Hypersensitivity,<br>Seizure) not reported to safety within the required<br>timeframe (within 24 hours of awareness for SAE;<br>within 72 hours of awareness for AESI) | Major / potentially critical |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | MRI or PET done before SV1 eligibility confirmed (lab and cog scales) | Major |
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | Tau PET scan conducted at Screening V3 with no confirmation of a positive amyloid result (either PET or CSF) from Screening Visits 1 or 2, or after meeting all other eligibility criteria, including MRI criteria, at Screening Visits 1 and 2. | Major |
| Study Procedures | Screening and baseline assessments not done, unless protocol allows them to be performed after day 1 | Major |
| Study Procedures | Infusion rate exceeds 100mL/hour | Major |
| Safety Monitoring | Dosing suspension decision has not been followed per protocol, MRI follow-up not performed correctly. | Major |
| Randomization | Screening window extended past 60 days without approval. | Minor (unless trending) |
| Visit schedule | Screening window extended beyond 90 days | Major |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| Study Procedures<br>(Study Procedures<br>(not safety not<br>efficacy related) | PET done prior to SV1 and MRI eligibility confirmed | Major |
| Blinding | First participant randomized at a site without signed Blind Maintenance Plan | Major |
| Visit schedule | Full visit not done NOTE: If MRI visit is skipped (either scheduled or unscheduled due to ARIA), see separate PD guidance for MRIs categorized under safety. | PD is MAJOR if any of the following apply: • > 2 consecutive visits are skipped • visit includes an infusion that was skipped for reasons other than ARIA (missed infusion reported separately) • visit includes CDR |
| Blinding | IP unblinded to blinded study team member or blinded site personnel | Major |
| Exclusion criteria | Vaccinations (including COVID-19 vaccines and boosters) within 5 days prior to randomization (Day 1). | Major |
| Concomitant<br>Medications | Vaccination < 5 days before a dosing visit and/or < 10 days after a dosing visit | Minor |
| Visit schedule<br>criteria | Subject missed 2 or more scheduled consecutive visits. | Major |
| Visit schedule<br>criteria | Failure to perform a required study visit that may affect subject safety or data integrity. | Major |
| Visit schedule<br>criteria | Failure to perform follow-up visit and/or End of Study Visit | Major |
| Visit schedule | Full study visit out of window (For full visits ONLY, this does not apply to individual procedures that may be done out of window) | Minor |

| Deviation<br>Category | Deviation Description | Severity<br>Classification |
|---|---|---|
| IP preparation | Site does not use the current weight, assessed at the current visit, for IP preparation | Major if the weight at the current visit is |
| | As this may be noted by the blinded team in the source documents (copies of weight communication to pharmacist and copy of weight at visit) or the unblinded team on the IP preparation documents both may report. This type of PD will need to be reconciled regularly to prevent duplication in the final log and to make sure none are missed. | the weight communicated dose preparation (regardless of under or overdose) Minor if the weight at the current visit is < 5 kg different from the weight communicated for the dose preparation |
| Other criteria | An unplanned unblinding of the subject or site to the subject's treatment information occurred during the study. | Major |

## **Certificate Of Completion**

Envelope Id: B3D41C54827343CAADEBFDDC529AE824

Subject: Complete with DocuSign: ENVISION SAP FINAL V1.0.pdf

Vendor Name: Source Envelope:

Document Pages: 52 Signatures: 4 Certificate Pages: 2 Initials: 0

AutoNav: Enabled

Envelopeld Stamping: Enabled

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

**Envelope Originator:** 

225 Binney St

Cambridge, MA 02142

IP Address:

#### Record Tracking

Status: Original

14 May 2024 | 09:22

Holder:

Location: DocuSign

#### Signer Events

Biostatistician

Biogen

Security Level: Email, Account Authentication

(None)

Signature

Signature Adoption: Pre-selected Style

Using IP Address:

**Timestamp** 

Sent: 14 May 2024 | 09:25 Viewed: 14 May 2024 | 09:46 Signed: 14 May 2024 | 09:47

## **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

Biostatistics

Biogen

Security Level: Email, Account Authentication

(None)

Signature Adoption: Pre-selected Style

Using IP Address:

Sent: 14 May 2024 | 09:47 Viewed: 14 May 2024 | 09:52 Signed: 14 May 2024 | 09:52

## **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

, Biostatistics

Biogen

Security Level: Email, Account Authentication (None)

Signature Adoption: Pre-selected Style Using IP Address:

Sent: 14 May 2024 | 09:52 Viewed: 14 May 2024 | 09:53 Signed: 14 May 2024 | 12:46

## **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign



Signature Adoption: Pre-selected Style Using IP Address:

Sent: 14 May 2024 | 12:46 Viewed: 14 May 2024 | 23:47 Signed: 14 May 2024 | 23:47

## Electronic Record and Signature Disclosure:

Not Offered via DocuSign

In Person Signer Events

Signature

**Timestamp** 

| Editor Delivery Events | Status | Timestamp |
|------------------------------|------------------|---------------------|
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 14 May 2024 09:25 |
| Certified Delivered | Security Checked | 14 May 2024 23:47 |
| Signing Complete | Security Checked | 14 May 2024 23:47 |
| Completed | Security Checked | 14 May 2024 23:47 |
| Payment Events | Status | Timestamps |